CLINICAL TRIAL: NCT02939118
Title: A One-Year, Multicenter, Observational, Follow-up Safety Study in Subjects Previously Implanted With VC-01™ Combination Product
Brief Title: One-Year Follow-up Safety Study in Subjects Previously Implanted With VC-01™
Status: Completed | Type: Observational
Sponsor: ViaCyte (Industry)
Responsible Party: Sponsor
Other Study IDs: VC01-201
Record Dates: First submitted 2016-10-18; First posted 2016-10-19 (Estimated); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this trial is to evaluate the long-term safety in subjects previously implanted with VC-01™ combination product.

ELIGIBILITY:
Inclusion Criteria:

* Previous implantation of VC-01™ combination product with subsequent explantation of all VC-01 units.

Exclusion Criteria:

* There are no exclusion criteria for this trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All subjects who have been exposed to implanted VC-01™ in any ViaCyte clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events reported during the study. | 12 months